CLINICAL TRIAL: NCT02995772
Title: Preoperative Neoadjuvant Hormonal Therapy and Neoadjuvant Chemotherapy for Stage IIIB and IV Breast Cancer Patients in Dharmais National Cancer Center Hospital, Indonesia
Brief Title: Neoadjuvant Hormonal Therapy Compared to Neoadjuvant Chemotherapy in Stage IIIB/C and IV Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dharmais National Cancer Center Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 049/PEP/08/2011
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Aromatase Inhibitors; Anastrozole; Tamoxifen; Fluorouracil; Doxorubicin; Cyclophosphamide; Letrozole; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant hormonal therapy (Active Comparator): Neoadjuvant hormonal therapy: Aromatase inhibitors (Arimidex, Femara, Aromasin), Tamoxifen, SOB and AI, SOB and Tamoxifen
  Interventions: Drug: Aromatase Inhibitors (Arimidex); Drug: Tamoxifen; Procedure: SOB; Drug: Aromatase Inhibitors (Femara); Drug: Aromatase Inhibitors (Aromasin)
- Neoadjuvant chemotherapy (Active Comparator): Neoadjuvant chemotherapy: FAC 6 cycles
  Interventions: Drug: FAC

INTERVENTIONS:
Drug: Aromatase Inhibitors (Arimidex) — Comparison of efficacy with chemotherapy
  Other Names: Anastrozole
  Arms: Neoadjuvant hormonal therapy
Drug: Tamoxifen — Comparison of efficacy with chemotherapy
  Other Names: Nolvadex; Soltamox
  Arms: Neoadjuvant hormonal therapy
Procedure: SOB — Comparison of efficacy with chemotherapy
  Other Names: Salpingo-oophorectomy Bilateral
  Arms: Neoadjuvant hormonal therapy
Drug: FAC — Comparison of efficacy with hormonal therapy
  Other Names: Fluorouracil, Adriamycin, Cytoxan
  Arms: Neoadjuvant chemotherapy
Drug: Aromatase Inhibitors (Femara) — Comparison of efficacy with chemotherapy
  Other Names: Letrozole
  Arms: Neoadjuvant hormonal therapy
Drug: Aromatase Inhibitors (Aromasin) — Comparison of efficacy with chemotherapy
  Other Names: Exemestane
  Arms: Neoadjuvant hormonal therapy

SUMMARY:
This study compared long term outcome of stage IIIB/C and IV breast cancer patients treated with neoadjuvant hormonal therapy (NAHT) and those treated with neoadjuvant chemotherapy (NACT)

DETAILED DESCRIPTION:
This study compared long term outcome of stage IIIB/C and IV breast cancer patients treated with neoadjuvant hormonal therapy (NAHT) and those treated with neoadjuvant chemotherapy (NACT) between 2011 and 2016.

The primary end points are overall survival (OS) and progression free survival (PFS) with Kaplan Meier.

This study was approved by Ethical Committee in Dharmais National Cancer Hospital.

ELIGIBILITY:
Inclusion Criteria:

* IIIB/C and IV stage of breast cancer
* received neoadjuvant hormonal therapy or neoadjuvant chemotherapy
* had first and second biopsy (surgery) within 6 months

Exclusion Criteria:

* had mastectomy before treatment
* pregnant
* disagree to enter the study
* had been given hormonal therapy or chemotherapy before study
* had contra-indication of SOB for pre-menopausal patients

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Overall survival | time from the date of pathological diagnosis until death from any cause and until minimum sample sizes are met and an average 3 years
  length of time from the date of pathological diagnosis until death from any cause

SECONDARY OUTCOMES:
Progressive free survival | time from after treatment until tumor progression or death from any cause and until minimum sample sizes are met and an average 3 years
  length of time from after treatment until tumor progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Ramadhan Karsono, Doctoral, Study Chair — Dharmais National Cancer Center Hospital
Locations (1):
- Dharmais National Cancer Center Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided on this yet

REFERENCES:
- [Result] Beatson GT. On the Treatment of Inoperable Cases of Carcinoma of the Mamma: Suggestions for a New Method of Treatment, with Illustrative Cases. Trans Med Chir Soc Edinb. 1896;15:153-179. No abstract available. PMID 29584099
- [Result] van de Vijver MJ, He YD, van't Veer LJ, Dai H, Hart AA, Voskuil DW, Schreiber GJ, Peterse JL, Roberts C, Marton MJ, Parrish M, Atsma D, Witteveen A, Glas A, Delahaye L, van der Velde T, Bartelink H, Rodenhuis S, Rutgers ET, Friend SH, Bernards R. A gene-expression signature as a predictor of survival in breast cancer. N Engl J Med. 2002 Dec 19;347(25):1999-2009. doi: 10.1056/NEJMoa021967. PMID 12490681
- [Result] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Result] Cardoso F, van't Veer LJ, Bogaerts J, Slaets L, Viale G, Delaloge S, Pierga JY, Brain E, Causeret S, DeLorenzi M, Glas AM, Golfinopoulos V, Goulioti T, Knox S, Matos E, Meulemans B, Neijenhuis PA, Nitz U, Passalacqua R, Ravdin P, Rubio IT, Saghatchian M, Smilde TJ, Sotiriou C, Stork L, Straehle C, Thomas G, Thompson AM, van der Hoeven JM, Vuylsteke P, Bernards R, Tryfonidis K, Rutgers E, Piccart M; MINDACT Investigators. 70-Gene Signature as an Aid to Treatment Decisions in Early-Stage Breast Cancer. N Engl J Med. 2016 Aug 25;375(8):717-29. doi: 10.1056/NEJMoa1602253. PMID 27557300
- [Result] Asad J, Jacobson AF, Estabrook A, Smith SR, Boolbol SK, Feldman SM, Osborne MP, Boachie-Adjei K, Twardzik W, Tartter PI. Does oncotype DX recurrence score affect the management of patients with early-stage breast cancer? Am J Surg. 2008 Oct;196(4):527-9. doi: 10.1016/j.amjsurg.2008.06.021. PMID 18809056
- [Result] Teshome M, Hunt KK. Neoadjuvant therapy in the treatment of breast cancer. Surg Oncol Clin N Am. 2014 Jul;23(3):505-23. doi: 10.1016/j.soc.2014.03.006. Epub 2014 Apr 24. PMID 24882348
- [Result] Mauriac L, MacGrogan G, Avril A, Durand M, Floquet A, Debled M, Dilhuydy JM, Bonichon F. Neoadjuvant chemotherapy for operable breast carcinoma larger than 3 cm: a unicentre randomized trial with a 124-month median follow-up. Institut Bergonie Bordeaux Groupe Sein (IBBGS). Ann Oncol. 1999 Jan;10(1):47-52. doi: 10.1023/a:1008337009350. PMID 10076721
- [Result] Chia YH, Ellis MJ, Ma CX. Neoadjuvant endocrine therapy in primary breast cancer: indications and use as a research tool. Br J Cancer. 2010 Sep 7;103(6):759-64. doi: 10.1038/sj.bjc.6605845. Epub 2010 Aug 10. PMID 20700118
- [Result] Bossuyt V, Provenzano E, Symmans WF, Boughey JC, Coles C, Curigliano G, Dixon JM, Esserman LJ, Fastner G, Kuehn T, Peintinger F, von Minckwitz G, White J, Yang W, Badve S, Denkert C, MacGrogan G, Penault-Llorca F, Viale G, Cameron D; Breast International Group-North American Breast Cancer Group (BIG-NABCG) collaboration. Recommendations for standardized pathological characterization of residual disease for neoadjuvant clinical trials of breast cancer by the BIG-NABCG collaboration. Ann Oncol. 2015 Jul;26(7):1280-91. doi: 10.1093/annonc/mdv161. Epub 2015 May 27. PMID 26019189
- [Result] Chuang E, Paul C, Flam A, McCarville K, Forst M, Shin S, Vahdat L, Swistel A, Simmons R, Osborne M. Breast cancer subtypes in Asian-Americans differ according to Asian ethnic group. J Immigr Minor Health. 2012 Oct;14(5):754-8. doi: 10.1007/s10903-012-9577-7. PMID 22286607
- [Result] Hammond ME, Hayes DF, Dowsett M, Allred DC, Hagerty KL, Badve S, Fitzgibbons PL, Francis G, Goldstein NS, Hayes M, Hicks DG, Lester S, Love R, Mangu PB, McShane L, Miller K, Osborne CK, Paik S, Perlmutter J, Rhodes A, Sasano H, Schwartz JN, Sweep FC, Taube S, Torlakovic EE, Valenstein P, Viale G, Visscher D, Wheeler T, Williams RB, Wittliff JL, Wolff AC; American Society of Clinical Oncology; College of American Pathologists. American Society of Clinical Oncology/College of American Pathologists guideline recommendations for immunohistochemical testing of estrogen and progesterone receptors in breast cancer (unabridged version). Arch Pathol Lab Med. 2010 Jul;134(7):e48-72. doi: 10.5858/134.7.e48. PMID 20586616
- [Result] Marcus DM, Switchenko JM, Prabhu R, O'Regan R, Zelnak A, Fasola C, Mister D, Torres MA. Neoadjuvant Hormonal Therapy is Associated with Comparable Outcomes to Neoadjuvant Chemotherapy in Post-Menopausal Women with Estrogen Receptor-Positive Breast Cancer. Front Oncol. 2013 Dec 27;3:317. doi: 10.3389/fonc.2013.00317. eCollection 2013. PMID 24409418
- [Result] Semiglazov VF, Semiglazov VV, Dashyan GA, Ziltsova EK, Ivanov VG, Bozhok AA, Melnikova OA, Paltuev RM, Kletzel A, Berstein LM. Phase 2 randomized trial of primary endocrine therapy versus chemotherapy in postmenopausal patients with estrogen receptor-positive breast cancer. Cancer. 2007 Jul 15;110(2):244-54. doi: 10.1002/cncr.22789. PMID 17538978
- [Result] Preece PE, Wood RA, Mackie CR, Cuschieri A. Tamoxifen as initial sole treatment of localised breast cancer in elderly women: a pilot study. Br Med J (Clin Res Ed). 1982 Mar 20;284(6319):869-70. doi: 10.1136/bmj.284.6319.869-a. No abstract available. PMID 6802332
- [Result] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Result] Schneeweiss A, Chia S, Hickish T, Harvey V, Eniu A, Hegg R, Tausch C, Seo JH, Tsai YF, Ratnayake J, McNally V, Ross G, Cortes J. Pertuzumab plus trastuzumab in combination with standard neoadjuvant anthracycline-containing and anthracycline-free chemotherapy regimens in patients with HER2-positive early breast cancer: a randomized phase II cardiac safety study (TRYPHAENA). Ann Oncol. 2013 Sep;24(9):2278-84. doi: 10.1093/annonc/mdt182. Epub 2013 May 22. PMID 23704196
- [Result] Hamy AS, Belin L, Bonsang-Kitzis H, Paquet C, Pierga JY, Lerebours F, Cottu P, Rouzier R, Savignoni A, Lae M, Reyal F. Pathological complete response and prognosis after neoadjuvant chemotherapy for HER2-positive breast cancers before and after trastuzumab era: results from a real-life cohort. Br J Cancer. 2016 Jan 12;114(1):44-52. doi: 10.1038/bjc.2015.426. Epub 2015 Dec 10. PMID 26657653
- [Result] Tashiro H, Nomura Y, Hisamatsu K. [A randomized trial of endocrine therapy, chemotherapy, and chemo-endocrine therapy in advanced breast cancer]. Gan To Kagaku Ryoho. 1990 Dec;17(12):2369-73. Japanese. PMID 2260873
- [Result] von Minckwitz G, Blohmer JU, Costa SD, Denkert C, Eidtmann H, Eiermann W, Gerber B, Hanusch C, Hilfrich J, Huober J, Jackisch C, Kaufmann M, Kummel S, Paepke S, Schneeweiss A, Untch M, Zahm DM, Mehta K, Loibl S. Response-guided neoadjuvant chemotherapy for breast cancer. J Clin Oncol. 2013 Oct 10;31(29):3623-30. doi: 10.1200/JCO.2012.45.0940. Epub 2013 Sep 3. PMID 24002511
- [Result] Abe O, Asaishi K, Izuo M, Enomoto K, Koyama H, Tominaga T, Nomura Y, Ohshima A, Aoki N, Tsukada T. Effects of medroxyprogesterone acetate therapy on advanced or recurrent breast cancer and its influences on blood coagulation and the fibrinolytic system. Surg Today. 1995;25(8):701-10. doi: 10.1007/BF00311486. PMID 8520164
- [Result] Saad ED, Katz A, Buyse M. Overall survival and post-progression survival in advanced breast cancer: a review of recent randomized clinical trials. J Clin Oncol. 2010 Apr 10;28(11):1958-62. doi: 10.1200/JCO.2009.25.5414. Epub 2010 Mar 1. PMID 20194852
- [Result] Wilcken N, Hornbuckle J, Ghersi D. Chemotherapy alone versus endocrine therapy alone for metastatic breast cancer. Cochrane Database Syst Rev. 2003;2003(2):CD002747. doi: 10.1002/14651858.CD002747. PMID 12804433
- [Result] Robertson JF, Todd JH, Ellis IO, Elston CW, Blamey RW. Comparison of mastectomy with tamoxifen for treating elderly patients with operable breast cancer. BMJ. 1988 Aug 20-27;297(6647):511-4. doi: 10.1136/bmj.297.6647.511. PMID 3139179
- [Result] Badwe R, Hawaldar R, Nair N, Kaushik R, Parmar V, Siddique S, Budrukkar A, Mittra I, Gupta S. Locoregional treatment versus no treatment of the primary tumour in metastatic breast cancer: an open-label randomised controlled trial. Lancet Oncol. 2015 Oct;16(13):1380-8. doi: 10.1016/S1470-2045(15)00135-7. Epub 2015 Sep 9. PMID 26363985